CLINICAL TRIAL: NCT04584970
Title: Evaluation of Virtual Reality Intervention After Pediatric Idiopathic Scoliosis Surgery to Reduce Postoperative Pain and Opioid Consumption
Brief Title: Virtual Reality After Pediatric Scoliosis Surgery
Acronym: VRAS-PS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0696
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-07

CONDITIONS: Scoliosis Idiopathic; Pain, Postoperative
Keywords: Virtual reality; Distraction methods; Idiopathic scoliosis; Postoperative pain; Pediatric surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual reality device (Experimental): Participants will be offered a virtual reality (VR) device for up to 30 minutes for two separate sessions on postoperative day 1. The device will be pre-loaded with a variety of vetted and screened age-appropriate games.
  Interventions: Device: Applied VR
- iPad device (Active Comparator): Participants will be offered an iPad device for up to 30 minutes for two separate sessions on postoperative day 1. The device will be pre-loaded with a variety of vetted and screened age-appropriate games.
  Interventions: Device: Apple iPad

INTERVENTIONS:
Device: Applied VR — The Applied VR device is a lightweight mobile virtual reality headset with embedded software, creating an immersive experience. The Applied VR is specifically designed for medical use.
  Arms: Virtual reality device
Device: Apple iPad — The Apple iPad is a tablet device controlled by touch screen with a variety of games and applications.
  Arms: iPad device

SUMMARY:
The purpose of this study is to evaluate the use of virtual reality after scoliosis surgery in pediatric patients.

DETAILED DESCRIPTION:
Purpose: To evaluate postoperative pain scores and postoperative opioid use in pediatric idiopathic scoliosis surgical patients using virtual reality (VR) as a method of immersive distraction compared with standard electronic use postoperatively.

Participants: Patients age 11-17 undergoing idiopathic scoliosis surgery on Enhanced Recovery After Surgery (ERAS) spine protocol at our institution.

Procedures (methods): Participants will be randomized to intervention arm (VR) or control arm (iPad). Baseline pain and anxiety scores will be assessed. On postoperative day 1, each patient will receive a visit by the research assistant who will assess pain scores, PCA use, etc. The intervention group will be offered a VR device for up to 30 minutes. The control group will be offered an iPad for up to 30 minutes. This visit will be performed twice on postoperative day 1. Follow up survey will be conducted at 48-72 hours and 7-10 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 11 - 17 years of age
* Patients undergoing idiopathic scoliosis surgery on Enhanced Recovery after Surgery (ERAS) spine protocol (which includes postoperative PCA)

Exclusion Criteria:

* Patient/caregiver refusal
* Patients with developmental delay
* Patients with seizure disorder
* Non-English-speaking patients
* Patients with daily opioid use >/= two weeks
* Patients with uncorrected visual or hearing impairment
* Patients admitted to pediatric intensive care unit on postoperative day #1

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Specht, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina (UNC) Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures, and appendices), will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to marley.lawrence@unchealth.unc.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following publication
Access Criteria: Researchers who present a methodologically sound proposal and return a signed data access agreement

REFERENCES:
- [Background] Arane K, Behboudi A, Goldman RD. Virtual reality for pain and anxiety management in children. Can Fam Physician. 2017 Dec;63(12):932-934. PMID 29237632
- [Background] Eijlers R, Legerstee JS, Dierckx B, Staals LM, Berghmans J, van der Schroeff MP, Wijnen RM, Utens EM. Development of a Virtual Reality Exposure Tool as Psychological Preparation for Elective Pediatric Day Care Surgery: Methodological Approach for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Sep 11;6(9):e174. doi: 10.2196/resprot.7617. PMID 28893727
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Piskorz J, Czub M. Effectiveness of a virtual reality intervention to minimize pediatric stress and pain intensity during venipuncture. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12201. Epub 2017 Nov 20. PMID 29155488
- [Background] Ryu JH, Park SJ, Park JW, Kim JW, Yoo HJ, Kim TW, Hong JS, Han SH. Randomized clinical trial of immersive virtual reality tour of the operating theatre in children before anaesthesia. Br J Surg. 2017 Nov;104(12):1628-1633. doi: 10.1002/bjs.10684. Epub 2017 Oct 4. PMID 28975600
- [Background] Won AS, Tataru CA, Cojocaru CM, Krane EJ, Bailenson JN, Niswonger S, Golianu B. Two Virtual Reality Pilot Studies for the Treatment of Pediatric CRPS. Pain Med. 2015 Aug;16(8):1644-7. doi: 10.1111/pme.12755. Epub 2015 Apr 30. No abstract available. PMID 25930099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality Device | iPad Device
Started | 11 | 12
Completed | 10 | 9
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Device | iPad Device | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Customized [Count of Participants; unit: Participants]
  Aged 11-14 | 6 | 7 | 13
  Aged 15-17 | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Via FACES Scale by Patient at Baseline
Description: All patients will be oriented to the Wong-Baker FACES Pain Rating scale preoperatively. This is a self-assessment scale; patients select a face that illustrates the pain they are experiencing. Scores 0-10, with 0=No hurt and 10=Hurts worst. Higher score indicates a worse outcome.
Time Frame: Recorded preoperatively as baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 11 | 12
score on a scale | 0.91 [0 to 4] | 0.92 [0 to 6]

2. Primary Outcome: Pain Scores Via FACES Scale by Patient at First Intervention Exposure T=0
Description: All patients will be oriented to the Wong-Baker FACES Pain Rating scale preoperatively. This is a self-assessment scale; patients select a face that illustrates the pain they are experiencing. Scores 0-10, with 0=No hurt and 10=Hurts worst. Higher score indicates a worse outcome. Assessed immediately prior to first intervention exposure (T=0 min) during 1 30-minute session on day 1 postoperatively.
Time Frame: Recorded immediately prior to intervention (T=0 min)
Population: Data not included for participants who withdrew from study
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 10 | 9
score on a scale | 5.00 [0 to 10] | 4.22 [0 to 8]

3. Primary Outcome: Pain Scores Via FACES Scale by Patient at First Intervention Exposure T=30
Description: All patients will be oriented to the Wong-Baker FACES Pain Rating scale preoperatively. This is a self-assessment scale; patients select a face that illustrates the pain they are experiencing. Scores 0-10, with 0=No hurt and 10=Hurts worst. Higher score indicates a worse outcome. Assessed immediately after first intervention exposure (T=30 min) following 1 30-minute session on day 1 postoperatively.
Time Frame: Recorded at end of intervention (T=30 minutes)
Population: Data not included for participants who withdrew from study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 10 | 9
score on a scale | 3.80 [0 to 8] | 3.55 [0 to 6]

4. Primary Outcome: Pain Scores Via FLACC Scale by Research Assistant at Baseline
Description: The Face, Legs, Arms, Cry and Consolability (FLACC) score will be measured by the trained research assistant. This is an observer assessment scale, with 5 categories (i.e., 'Face', with 0=No particular expression or smile, 1=Occasional grimace or frown, 2=Frequent to constant quivering chin, clenched jaw). Scores 0-2 in each category, for total scores 0-10, with 0=No observed pain and 10=Most observed pain. Higher score indicates a worse outcome.
Time Frame: Recorded preoperatively as baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 11 | 12
score on a scale | 0 (0) | 1.5 (3.12)

5. Primary Outcome: Pain Scores Via FLACC Scale by Research Assistant at First Intervention Exposure T=0
Description: The Face, Legs, Arms, Cry and Consolability (FLACC) score will be measured by the trained research assistant. This is an observer assessment scale, with 5 categories (i.e., 'Face', with 0=No particular expression or smile, 1=Occasional grimace or frown, 2=Frequent to constant quivering chin, clenched jaw). Scores 0-2 in each category, for total scores 0-10, with 0=No observed pain and 10=Most observed pain. Higher score indicates a worse outcome. Assessed immediately prior to first intervention exposure (T=0 min) during 1 30-minute session on day 1 postoperatively.
Time Frame: Recorded immediately prior to intervention (T=0 minutes)
Population: Data not included for participants who withdrew from study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 10 | 9
score on a scale | 0.60 (1.07) | 0.33 (0.71)

6. Primary Outcome: Pain Scores Via FLACC Scale by Research Assistant at First Intervention Exposure T=10
Description: The Face, Legs, Arms, Cry and Consolability (FLACC) score will be measured by the trained research assistant. This is an observer assessment scale, with 5 categories (i.e., 'Face', with 0=No particular expression or smile, 1=Occasional grimace or frown, 2=Frequent to constant quivering chin, clenched jaw). Scores 0-2 in each category, for total scores 0-10, with 0=No observed pain and 10=Most observed pain. Higher score indicates a worse outcome. Assessed immediately during first intervention exposure (T=10 min) during 1 30-minute session on day 1 postoperatively.
Time Frame: Recorded at the 10 minute mark (T=10 minutes)
Population: Data not included for participants who withdrew from study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 10 | 9
score on a scale | 0 (0) | 0.44 (1.33)

7. Primary Outcome: Pain Scores Via FLACC Scale by Research Assistant at First Intervention Exposure T=30
Description: The Face, Legs, Arms, Cry and Consolability (FLACC) score will be measured by the trained research assistant. This is an observer assessment scale, with 5 categories (i.e., 'Face', with 0=No particular expression or smile, 1=Occasional grimace or frown, 2=Frequent to constant quivering chin, clenched jaw). Scores 0-2 in each category, for total scores 0-10, with 0=No observed pain and 10=Most observed pain. Higher score indicates a worse outcome. Participants were allowed to play/interact with intervention for up to 30 minutes. Assessed immediately following first intervention exposure (T=30 min) following 1 30-minute session on day 1 postoperatively.
Time Frame: Recorded at end of intervention (T=30 minutes)
Population: Data not included for participants who withdrew from study. Data are included for those participants who interacted with the intervention for the full 30-minute time limit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 5 | 7
score on a scale | 0 (0) | 0 (0)

8. Primary Outcome: Opioid PCA Use at T=-60-0
Description: Opioid use via Patient-Controlled Analgesia (PCA) pump in mcg or mg as appropriate. PCA use will be converted to morphine equivalents at time of data entry. A higher number indicates more opioid used during the time interval. Higher number indicates a worse outcome.
Time Frame: Recorded for the hour prior to intervention (T=-60-0 minutes)
Population: PCA pumps were no longer in use by the time the study intervention was employed; therefore, these data were not collected.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Opioid PCA Use at T=0-30
Description: Opioid use via PCA pump in mcg or mg as appropriate. PCA use will be converted to morphine equivalents at time of data entry. A higher number indicates more opioid used during the time interval. Higher number indicates a worse outcome.
Time Frame: Recorded during intervention (T=0-30 minutes)
Population: as for outcome 8
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Opioid PCA Use at T=30-90
Description: as for outcome 9
Time Frame: Recorded one hour after intervention is complete (T=30-90 minutes)
Population: as for outcome 8
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Total Opioid Dose (in Milligram Morphine Equivalents)
Description: The amount of opioids used by the patient will be recorded in all subjects and converted into milligram morphine equivalents based on chart reviews. This collection method was added to replace PCA pump usage unavailability.
Time Frame: From anesthesia end through hospital discharge, a total of approximately 2 days
Population: Data not included for participants who withdrew from study.
Measure: Mean (Standard Deviation); unit: (mg) morphine equivalents
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 10 | 9
(mg) morphine equivalents | 4.74 (1.19) | 5.27 (1.52)

12. Secondary Outcome: Electronic Device Use
Description: VR device or iPad use in minutes. Minimal 0 minutes, maximum 60 minutes (30 minutes x 2 sessions). A higher number indicates more electronic device use, which is neither a better or worse outcome, but rather provides information about whether devices were used for the full allotted time or not.
Time Frame: Assessed at time of intervention on postoperative day #1
Population: Data not included for participants who withdrew from study and an additional 2 participants for whom data were inadvertently not recorded.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 9 | 8
minutes | 20.33 (7.58) | 26.38 (4.44)

13. Secondary Outcome: Baseline Anxiety Score Via STAI Short Form Baseline Anxiety Score Via STAI Short Form
Description: The State-Trait Anxiety Inventory (STAI) Short Form scoring tool is a self-report questionnaire. It contains 6 statements (i.e., 'I feel calm', with 1=Not at all, 2=Somewhat, 3=Moderately, 4=Very much). Scores range from 6-24, with 6 signifying no anxiety and 24 points signifying the highest level of anxiety. Higher score indicates a worse outcome.
Time Frame: Recorded preoperatively as baseline
Population: Data were not collected for 1 participant in the iPad device group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 11 | 11
score on a scale | 11.64 (3.29) | 13.27 (4.86)

14. Secondary Outcome: Postoperative Behavioral Changes Via PHBQ-AS Form at 48-72 Hours
Description: A follow up survey will be given using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS) form via a phone call, email or in person from a member of the research team. There are 11 items on a five-point scale (i.e., 1=Much less than before, 5=Much more than before). Total scores 11-55, with higher scores indicating more negative behavioral changes. Higher score indicates a worse outcome.
Time Frame: At approximately 48-72 hours postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Postoperative Behavioral Changes Via PHBQ-AS Form at 7-10 Days
Description: as for outcome 14
Time Frame: At approximately 7-10 days postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Patient Satisfaction at 48-72 Hours
Description: To assess patient satisfaction, qualitative satisfaction will be documented. Patient satisfaction and overall experience are commonly linked to pain experienced during a hospitalization, and as a result, satisfaction with the use of VR as a method of pain control will be one of the outcomes. Patients will simply be asked by the researcher assistant, qualitatively, how satisfied they were with their experience with the device, and their comments will be recorded. Collected answers will be divided into positive and negative comments, and any emerging themes will be identified.
Time Frame: At approximately 48-72 hours postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Patient Satisfaction at 7-10 Days
Description: as for outcome 16
Time Frame: At approximately 7-10 days postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Caregiver Satisfaction at 48-72 Hours
Description: To assess caregiver satisfaction, qualitative satisfaction will be documented. Patient and caregiver satisfaction and overall experience are commonly linked to pain experienced during a hospitalization, and as a result, satisfaction with the use of VR as a method of pain control will be one of the outcomes. Caregivers will simply be asked by the researcher assistant, qualitatively, how satisfied they were with their child's experience with the device, and their comments will be recorded. Collected answers will be divided into positive and negative comments, and any emerging themes will be identified.
Time Frame: At approximately 48-72 hours postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Caregiver Satisfaction at 7-10 Days
Description: as for outcome 18
Time Frame: At approximately 7-10 days postoperatively
Population: Due to COVID-19, all questionnaires were sent via email; however, no responses were received.
Arm/Group | Virtual Reality Device | iPad Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During two 30-minute post-operative intervention visits, a total of approximately 1 hour.
Arm/Group | Virtual Reality Device | iPad Device
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04584970/Prot_SAP_000.pdf